CLINICAL TRIAL: NCT06022926
Title: Effects of Patient Warming With Electric Blanket on Intraoperative Hemodynamics; Postoperative Nausea, Vomiting, Chills, Agitation and Pain in Laparoscopic Cholecystectomy Operation
Brief Title: Investigation of the Intraoperative and Postoperative Effects of Warming Patients in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Anesthesiology and Reanimation Spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11.25.2022/235
Record Dates: First submitted 2023-08-15; First posted 2023-09-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Patients warmed with electric blankets (Active Comparator): * Patients will be provided with electric blankets from the beginning to the end of the operation (approximately 1 hour)
  * all patients will receive standard general anesthesia
  * each patient will undergo tympanic temperature measurement immediately before induction of general anesthesia, 20 minutes after induction of anesthesia, immediately after extubation and during exit from the postanesthesia recovery unit.
  * the same electric blanket was used for this group of patients
  * each time the electric blankets were set to 38 degrees and the blankets were preheated to 38 degrees approximately 30 minutes before the patients were placed on the operating table.
  * heat measurements will be made with the same tympanic heat meter device
  Interventions: Procedure: warmed with electric blankets
- Group 2: Control group (patients without warming) (Other): * no electric blanket will be used, and no heating will be applied to this group of patients.
  * all patients will receive standard general anesthesia
  * all patients will undergo electrocardiogram, peripheral oxygen saturation by pulse oximetry, non-invasive blood pressure monitoring by automatic pneumatic manometer
  * mean arterial pressure, intraoperative opioid consumption, nausea-vomiting, agitation, tremor and pain assessment will be performed on each patient immediately before induction of general anesthesia, 20 minutes after induction of anesthesia, immediately after extubation and during discharge from the postanesthesia recovery unit.
  * temperature measurements will be performed with the same tympanic thermometer device
  Interventions: Other: patients without warming

INTERVENTIONS:
Procedure: warmed with electric blankets — warmed with electric blankets
  Arms: Group 1: Patients warmed with electric blankets
Other: patients without warming — patients without warming: no electric blanket will be used, and no heating will be applied to this group of patients.
  Arms: Group 2: Control group (patients without warming)

SUMMARY:
In our study, the investigators will investigate the effects of electric blanket heating on intraoperative hemodynamics, postoperative nausea, vomiting, shivering, agitation and pain in patients undergoing laparoscopic cholecystectomy under general anesthesia.

DETAILED DESCRIPTION:
Group 1: Patients warmed with electric blankets

* Patients will be provided with electric blankets from the beginning to the end of the operation (approximately 1 hour)
* all patients will receive standard general anesthesia
* all patients will undergo electrocardiogram, peripheral oxygen saturation by pulse oximetry, non-invasive blood pressure monitoring by automatic pneumatic manometer.
* each patient will undergo tympanic temperature measurement immediately before induction of general anesthesia, 20 minutes after induction of anesthesia, immediately after extubation and during exit from the postanesthesia recovery unit.
* mean arterial pressure, intraoperative opioid consumption, nausea-vomiting, agitation, tremor and pain assessment will be performed on each patient immediately before induction of general anesthesia, 20 minutes after induction of anesthesia, immediately after extubation and during discharge from the postanesthesia recovery unit.
* the same electric blanket was used for this group of patients
* each time the electric blankets were set to 38 degrees and the blankets were preheated to 38 degrees approximately 30 minutes before the patients were placed on the operating table.
* heat measurements will be made with the same tympanic heat meter device
* heat measurements will be made by a blind anesthesiologist with at least 5 years of experience
* Postoperative evaluations of the patients will be performed face to face.
* patients will be warmed only during the time they are on the operating table
* This study was followed up in the operating room and post-anesthesia recovery unit in the operating room.

Group 2: Control group (patients without warming): no electric blanket will be used, and no heating will be applied to this group of patients.

* all patients will receive standard general anesthesia.
* all patients will undergo electrocardiogram, peripheral oxygen saturation by pulse oximetry, non-invasive blood pressure monitoring by automatic pneumatic manometer.
* each patient will undergo tympanic temperature measurement immediately before induction of general anesthesia, 20 minutes after induction of anesthesia, immediately after extubation and during exit from the postanesthesia recovery unit.
* mean arterial pressure, intraoperative opioid consumption, nausea-vomiting, agitation, tremor and pain assessment will be performed on each patient immediately before induction of general anesthesia, 20 minutes after induction of anesthesia, immediately after extubation and during discharge from the postanesthesia recovery unit.
* temperature measurements will be performed with the same tympanic thermometer device
* heat measurements will be made by a blind anesthesiologist with at least 5 years of experience
* Postoperative evaluations of the patients will be performed face to face.
* This study was followed up in the operating room and post-anesthesia recovery unit in the operating room.

Statistical methods / analysis: G-Power version 3.1.9.4 (University Kiel, Germany) was used to calculate the sample size. Two-tailed alpha error was 0.05, power as 0.80 and effect size as 0.5, and according to a previous study (Comparison of different end-tidal carbon dioxide levels in preventing postoperative nausea and vomiting in gynaecological patients undergoing laparoscopic surgery. Doi: 10.1080/01443615.2020.1789961.) allocation ratio was accepted as N2/N1:1. The minimum number of patients to be included in the study was calculated as 128.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy operation will be
* To be between 18-65 years old.
* Being American Society of Anesthesiologists (ASA) Classification I-II.

Exclusion Criteria:

* Preoperative body temperature >37.5°C or <36°C.
* Impaired temperature regulation such as systemic infection, mental retardation, isolated head trauma or brain injury.
* Receiving a medication that affects thermoregulation.
* Being American Society of Anesthesiologists (ASA) Classification >III.

Ages: 18 Days to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Agitation assessment | Will be assessed from immediately after extubation until transfer from the recovery room to the ward.
  Agitation assessment with Richmond Agitation Sedation Scale (RASS). The Richmond Agitation Sedation Scale (RASS) is a 10-point scale ranging from -5 to +4.Levels -1 to -5 denote 5 levels of sedation, starting with "awakens to voice" and ending with "unarousable." Levels +1 to +4 describe increasing levels of agitation. The lowest level of agitation starts with apprehension and anxiety, and peaks at combative and violent. RASS level 0 is "alert and calm.

SECONDARY OUTCOMES:
Pain assessment | Within 30 minutes from the time the patient was extubated to the time of extubation from the postoperative recovery unit to the ward.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
post-operative tremor | Within 30 minutes from the time the patient was extubated to the time of extubation from the postoperative recovery unit to the ward.
  The evaluation will be made according to this rating:
  Grade 1: no tremor Grade 2: mild tremor with mild facial and cervical muscle contraction Grade 3: moderate tremor with obvious tremor of the head and neck, shoulders and/or extremities Grade 4: severe tremor consisting of an obvious tremor all over the body
Amount of fentanyl consumed intraoperatively | during surgery]
  micrograms of fentanyl consumed
Average blood pressure | Assessments will be performed at 0 minutes immediately before induction of anesthesia, 20 minutes after induction, immediately after extubation and 20 minutes in the recovery unit after anesthesia.
  Blood pressure will be measured with a non-invasive automatic pneumatic cuff in the operating theatre.
Heart rate | Assessments will be performed at 0 minutes immediately before induction of anesthesia, 20 minutes after induction, immediately after extubation and 20 minutes in the recovery unit after anesthesia.
  the measurement will be obtained by electrocardiographic monitoring
nausea-vomiting | The evaluation will be performed at postoperative 0th hour, 2nd hour, 6th hour and 24th hour.
  -Postoperative nausea and vomiting will be assessed using a 100 mm VAS:
  1- severe nausea (VAS>70 mm), 2- moderate nausea (50<VAS<70 mm), 3- mild nausea (VAS <50 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Cem K. Kaçar, Assoc.Prof, Study Director — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanaka N, Ohno Y, Hori M, Utada M, Ito K, Suzuki T. A randomised controlled trial of the resistive heating blanket versus the convective warming system for preventing hypothermia during major abdominal surgery. J Perioper Pract. 2013 Apr;23(4):82-6. doi: 10.1177/175045891302300404. PMID 23691884
- [Derived] Dedeoglu A, Acil F, Andic O, Ozkilic M. Effect of Intraoperative Active Warming Initiated at Anesthesia Induction on Core Temperature, Postoperative Pain and Agitation in Laparoscopic Cholecystectomy: A Randomized Controlled Trial. Medicina (Kaunas). 2026 Jan 15;62(1):175. doi: 10.3390/medicina62010175. PMID 41597461